CLINICAL TRIAL: NCT02484157
Title: Comparison of Activated Coagulation Time Between Hemochron Jr and ACT Plus During Cardiac Surgery for Patient Using Acute Normovolemic Hemodilution
Brief Title: Comparison of ACT Between Hemochron Jr and ACT Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2012-I0814
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2012-12

CONDITIONS: Cardiac Disease
Keywords: Whole Blood Coagulation Time; cardiac surgery
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient (Experimental): Patients were checked activated coagulation time by both Hemochron Jr and ACT Plus during cardiac surgery with heparin administration.
  Interventions: Device: Hemochron; Device: ACT Plus

INTERVENTIONS:
Device: Hemochron — Activated coagulation time was checked serially by Hemochron Jr.
Device: ACT Plus — Activated coagulation time was checked serially by ACT Plus.

SUMMARY:
This study aimed to compare 2 activated clotting time analysers (Hemochron Jr vs. ACT Plus).

DETAILED DESCRIPTION:
Measurement of activated clotting time (ACT) is a standard method for anticoagulation monitoring. Especially in cardiac surgery, heparin is usually used as anticoagulant and protamine is used to reverse anticoagulation effect at the end of surgery. ACT method defines the time until a clot is formed in a test tube after triggering of internal pathway coagulation using blood activating agents (eg. kaolin).

Acute normovolemic hemodilution (ANH) consists of withdrawing patient's blood volume early in the operative period and concurrent infusion of crystalloid or colloid to maintain intravascular volume, and is used in cardiac surgery. ANH is known to affect hemostasis in some studies.

Assuming that accurate monitoring of coagulation therapy is important to prevent both thrombotic and hemorrhagic complications, we compared ACT results from 2 analysers (Hemochron Jr and ACT Plus) in patients undergoing cardiac surgery using ANH.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent cardiac surgery with heparin administration.

Exclusion Criteria:

* Preoperative hemoglobin under 11g/dL
* Weight under 40kg
* Preoperative coagulopathy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Comparison of activated coagulation time between Hemochron Jr and ACT Plus | During cardiac surgeris (within 8 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Soo Kyung Lee, MD, Study Chair — Hallym University Medical Center
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Svenmarker S, Appelblad M, Jansson E, Haggmark S. Measurement of the activated clotting time during cardiopulmonary bypass: differences between Hemotec ACT and Hemochron Jr apparatus. Perfusion. 2004;19(5):289-94. doi: 10.1191/0267659104pf755oa. PMID 15506033
- [Background] Chia S, Van Cott EM, Raffel OC, Jang IK. Comparison of activated clotting times obtained using Hemochron and Medtronic analysers in patients receiving anti-thrombin therapy during cardiac catheterisation. Thromb Haemost. 2009 Mar;101(3):535-40. PMID 19277416
- [Background] Bosch YP, Weerwind PW, Nelemans PJ, Maessen JG, Mochtar B. An evaluation of factors affecting activated coagulation time. J Cardiothorac Vasc Anesth. 2012 Aug;26(4):563-8. doi: 10.1053/j.jvca.2012.03.011. Epub 2012 Apr 24. PMID 22534410
- [Background] Dalbert S, Ganter MT, Furrer L, Klaghofer R, Zollinger A, Hofer CK. Effects of heparin, haemodilution and aprotinin on kaolin-based activated clotting time: in vitro comparison of two different point of care devices. Acta Anaesthesiol Scand. 2006 Apr;50(4):461-8. doi: 10.1111/j.1399-6576.2006.00990.x. PMID 16548858